CLINICAL TRIAL: NCT07205042
Title: A Randomized Controlled Trial of a 12-Week Walking Program on Metabolic and Psychophysiological Outcomes in Women With Hypothyroidism
Brief Title: Walking for Hypothyroidism Trial (WHT)
Acronym: WHT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Advanced Education & Research Center (Other)
Responsible Party: Principal Investigator, Shamoon Noushad, Professor, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AEIRC-KU-2025-WHT01
Record Dates: First submitted 2025-09-13; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hypothyroidism
Keywords: Walking; Aerobic Exercise; Basal Metabolic Rate; Heart Rate Variability; Salivary Cortisol
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into two arms: (1) a 12-week supervised walking program and (2) a control group maintaining usual activity. Each group is followed in parallel for the full duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The walking program cannot be blinded to participants or exercise staff. However, outcome assessors (BMR testing, HRV analysis, cortisol assays) and statisticians will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking Intervention (Experimental): Participants will undergo a supervised walking program consisting of 30 minutes per session, 5 sessions per week, for 12 weeks. Exercise intensity will be maintained at 55-65% of age-predicted maximum heart rate, monitored by chest strap or optical heart rate sensors. Sessions will be supervised by an exercise physiologist, with adherence tracked through session logs and heart rate recordings. Participants will continue their usual levothyroxine regimen but will not initiate any new structured exercise program during the study period.
  Interventions: Behavioral: Supervised Walking Program
- Control (Usual Activity) (No Intervention): Participants will continue their usual daily routines without a prescribed exercise program. They will be instructed not to initiate any new structured exercise during the study. Weekly check-ins will be conducted to record incidental activity and monitor health status. At study completion, control participants will be offered the walking program.

INTERVENTIONS:
Behavioral: Supervised Walking Program — A structured walking program consisting of 30 minutes per session, 5 sessions per week, for 12 weeks at 55-65% of age-predicted maximum heart rate. Sessions will be supervised by an exercise physiologist, with adherence monitored by heart rate tracking and attendance logs. Participants will continue their standard levothyroxine treatment but will not begin any new structured exercise programs.
  Other Names: Aerobic walking, treadmill walking, moderate-intensity exercise
  Arms: Walking Intervention

SUMMARY:
Women with hypothyroidism often report persistent fatigue, weight gain, autonomic dysregulation, and stress despite stable levothyroxine therapy. This single-center, parallel-group RCT will test whether a structured, supervised 12-week walking program improves basal metabolic rate (BMR) and psychophysiological outcomes compared with usual activity. One hundred twenty women aged 35-55 with stable primary hypothyroidism will be randomized 1:1 to intervention or control.

DETAILED DESCRIPTION:
This trial evaluates a pragmatic, low-cost aerobic intervention-walking 30 minutes/day, 5 days/week at 55-65% HRmax for 12 weeks-as an adjunct to standard pharmacotherapy. Expected benefits: ↑BMR, ↑HRV, ↓cortisol, ↓fatigue, and improved mood. Outcome assessors/statisticians are masked; allocation is concealed. Safety monitoring covers musculoskeletal events, cardiovascular symptoms, and thyroid-related issues.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 35-55 years
* Primary hypothyroidism with documented prior TSH >4.5 mIU/L
* Stable levothyroxine dose for at least 6 months
* Sedentary lifestyle (<150 minutes of moderate-vigorous activity per week)
* BMI between 20-35 kg/m²
* Able to walk unaided
* Willing and able to provide written informed consent

Exclusion Criteria:

* Pregnant or lactating, or planning pregnancy during the study period
* Use of beta-blockers, systemic corticosteroids, or medications significantly affecting heart rate, HRV, or metabolism
* Uncontrolled hypertension, insulin-dependent diabetes, symptomatic cardiovascular disease, or orthopedic conditions limiting walking
* Major psychiatric hospitalization in the past 12 months
* Participation in another interventional trial within the past 30 days

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Basal Metabolic Rate | Basal metabolic rate (BMR) measured via indirect calorimetry under standardized conditions (fasted, thermoneutral room, supine rest ≥30 minutes). The primary analysis will compare change from baseline to 12 weeks between intervention and control groups.
  Baseline (Week 0) and Week 12

SECONDARY OUTCOMES:
Change in Heart Rate Variability | Baseline (Week 0) and Week 12
  Resting 5-minute ECG with paced breathing; RMSSD calculated after artifact correction.
Change in Heart Rate Variability | Baseline (Week 0) and Week 12
  Resting 5-minute ECG with paced breathing; SDNN calculated after artifact correction.
Change in Morning Salivary Cortisol | Baseline (Week 0) and Week 12
  Triplicate saliva samples collected at 08:00 h on two weekdays, pooled and assayed via ELISA.
Change in Fatigue Severity Scale | Baseline (Week 0) and Week 12
  Self-reported validated questionnaire; higher scores = greater fatigue.
Change in Hospital Anxiety and Depression Scale | Baseline (Week 0) and Week 12
  Self-reported validated questionnaire; higher scores = greater anxiety or depression symptoms.

OTHER OUTCOMES:
Adherence to Walking Program | Weekly throughout the 12-week intervention period
  Percentage of prescribed sessions completed, based on attendance logs and heart rate monitor data.
Adverse Events | From Week 1 through Week 12 (study intervention period)
  Weekly surveillance of adverse events, classified by type, severity, and seriousness.

CONTACTS AND LOCATIONS:
Overall Officials: Sadaf Ahmed, Ph.D., Principal Investigator — University of Karachi
Locations (1):
- University of Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected during this study will not be made publicly available due to ethical and privacy considerations. Summary results will be disseminated in scientific publications and presentations.

REFERENCES:
- [Background] Sundus H, Khan SA, Zaidi S, Chhabra C, Ahmad I, Khan H. Effect of long-term exercise-based interventions on thyroid function in hypothyroidism: A systematic review and meta-analysis of randomized controlled trials. Complement Ther Med. 2025 Sep;92:103196. doi: 10.1016/j.ctim.2025.103196. Epub 2025 May 28. PMID 40446861
- [Background] Dunabeitia I, Gonzalez-Devesa D, Varela-Martinez S, Diz-Gomez JC, Ayan-Perez C. Effect of physical exercise in people with hypothyroidism: systematic review and meta-analysis. Scand J Clin Lab Invest. 2023 Dec;83(8):523-532. doi: 10.1080/00365513.2023.2286651. Epub 2024 Jan 24. PMID 37999992
- [Background] Mathene Koteles E, Rafael B, Korom A, Vagvolgyi A, Abraham JE, Domjan A, Szucs M, Nemes A, Barnai M, Lengyel C, Kosa I. Physiological and psychological effects of a 12-week home-based telemonitored training in metabolic syndrome. Front Cardiovasc Med. 2023 Jan 10;9:1075361. doi: 10.3389/fcvm.2022.1075361. eCollection 2022. PMID 36704473
- [Background] Ahmad AM, Serry ZH, Abd Elghaffar HA, Ghazi HA, El Gayar SL. Effects of aerobic, resistance, and combined training on thyroid function and quality of life in hypothyroidism. A randomized controlled trial. Complement Ther Clin Pract. 2023 Nov;53:101795. doi: 10.1016/j.ctcp.2023.101795. Epub 2023 Aug 22. PMID 37659172